CLINICAL TRIAL: NCT04348903
Title: Effect of Virtual Reality Distraction Versus Positive Pre-Visit Imagery Intervention on Children's Dental Fear and Anxiety : Implications for Evidence-Based Practice
Brief Title: Virtual Reality Distraction Versus Positive Pre-Visit Imagery Intervention on Children's Dental Fear and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2113042020
Record Dates: First submitted 2020-04-03; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Nurse's Role
Keywords: Virtual Reality; Positive Pre-visit Imagery; Dental Fear; Dental anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Experimental): Virtual reality refers to a human-computer interface that completely immerse the child in a simulated environment. It integrates multiple perceptual senses including; the visual, auditory and kinaesthetic stimulation modalities. Virtual reality diverts children's attention away from the negative feelings associated with unpleasant experience.
  Interventions: Behavioral: Virtual Reality Distraction
- Positive Pre-Visit Imagery Intervention (Experimental): Positive pre-visit imagery is one of the superior cognitive- behavioral interventions. It is kind of psychological preparation that is designed to provide children with a step-by-step explanation of the dental local anaesthesia injection in an attractive approach
  Interventions: Behavioral: Positive Pre-Visit Imagery Intervention

INTERVENTIONS:
Behavioral: Virtual Reality Distraction — The researchers will prepare the VR device. The researches will explain the aim of using VR and adopt tell-show-do technique in introducing VR Glasses. Once VR device headset will be adapted to the child's head size and adjusted in front of his/her eyes, the selected 3D cartoon movie will be played in the waiting room and throughout the procedure of dental LA injection. After ensuring that the child is fully immersed in the cartoon movie, a needle of local anesthetic agent will be prepared and injected after explanation of the procedure.
  Arms: Virtual Reality Distraction
Behavioral: Positive Pre-Visit Imagery Intervention — Short narrative visual information regarding the dental chair, environment and equipment will be provided. It will be done through showing children an interactive book that contained photographs of A4 size, depicting three children model aged 4 - 6 years who are smiling while sitting in the dental chair and cooperative with the dentist. Benefit of LA in alleviating pain will be explained. The researchers also will explore the children's reflection of the children model and allow them ask questions relevant to LA injection.
  Arms: Positive Pre-Visit Imagery Intervention

SUMMARY:
Aim

This study aimed to determine the effect of virtual reality distraction versus positive pre-visit imagery intervention on children's dental fear and anxiety during local anaesthesia injection.

Research Hypotheses

1. Children who receive Virtual reality distraction or Positive pre-visit imagery intervention exhibit less dental fear and anxiety levels during LA injection than those who do not.
2. Children who receive Virtual reality distraction exhibit less dental fear and anxiety levels during LA injection than those who receive Positive pre-visit imagery intervention.

DETAILED DESCRIPTION:
Promoting children's health is a crucial nursing role. Dental health and psychological well-being are basic components of the health promotion for young children. Dental procedures especially local anesthesia injection is one of the most unpleasant experiences for young children. Dental Fear and Anxiety are considered pervasive psychological problems accompanied with strong negative feelings among a large portion of young children. Basically, dental fear and anxiety have been reported as one of the most important reasons for avoidance of dental treatments among young children, thereby results in an adverse effects on their oral and psychological health.

Nurses face a great challenge to minimize dental fear and anxiety and stabilize young children psychologically during restorative dental procedures. Such stabilization is the cornerstone of successful local anaesthesia injection and facilitating dentist's mission.

Virtual reality refers to a human-computer interface that completely immerse the child in a simulated environment. It integrates multiple perceptual senses including; the visual, auditory and kinaesthetic stimulation modalities. Virtual reality diverts children's attention away from the negative feelings associated with unpleasant experience.

Positive pre-visit imagery is one of the superior cognitive- behavioral interventions. It is kind of psychological preparation that is designed to provide children with a step-by-step explanation of the dental local anaesthesia injection in an attractive approach. It helps them to anticipate, deal with, and be empowered to gain mastery over the events they will experience. It also plays a role in counteracting the distorted beliefs that invading the children's conscious awareness.

ELIGIBILITY:
Inclusion Criteria

* Age ranged from 4- 6 years.
* Had a previous experience of dental local anaesthesia injection.
* Had carious mandibular primary molar and planned for restorative dental treatment.

Exclusion Criteria:

* Age more than 6 years.
* visual or auditory deficits.
* chronic or mental disabilities that affect their understanding.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2020-04-16 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Dental Local Anaesthesia Injection Fear Scale | 10 minutes
  This was scale developed by the researchers after thorough review of related literature to measure children's dental fear during dental local anaethesia injection (Riba et al., 2017 & Malhotra et al., 2018). It consisted of 15 items that emphasized on observing children's fear behavioral response. The scale comprises of two main categories including avoidant behaviors such as refuses to leave caregiver, sits on the dental chair or opens mouth in addition to over-exaggerated behaviors, such as attempts to dislodge syringe, kicks the doctor and leaves the chair. Each item was measured on a two-points Likert scale ranged from zero "behavior is not present" to one "behavior is present".
Venham's Dental Clinical Anxiety Rating Scale | 10 minutes
  This scale was developed by Venham and Kremer (1979) to quantify the anxious behaviors of 4-6 years-old children during situational dental anxiety. It is consisted of 6 items that were rated from relaxed to out of contact and were given numeric digit from zero to five respectively as follows: The scale was reliable and valid and can be easily integrated in clinical or research activities. Its content validity was 0.91 and a test-retest reliability revealed to be 0.93.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addicks SH, McNeil DW, Randall CL, Goddard A, Romito LM, Sirbu C, Kaushal G, Metzger A, Weaver BD. Dental Care-Related Fear and Anxiety: Distress Tolerance as a Possible Mechanism. JDR Clin Trans Res. 2017 Jul;2(3):304-311. doi: 10.1177/2380084417691962. Epub 2017 Feb 9. PMID 28879250
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Fox C, Newton JT. A controlled trial of the impact of exposure to positive images of dentistry on anticipatory dental fear in children. Community Dent Oral Epidemiol. 2006 Dec;34(6):455-9. doi: 10.1111/j.1600-0528.2006.00303.x. PMID 17092274
- [Background] Gangwal RR, Rameshchandra Badjatia S, Harish Dave B. Effect of Exposure to Positive Images of Dentistry on Dental Anxiety among 7 to 12 Years Old Children. Int J Clin Pediatr Dent. 2014 Sep-Dec;7(3):176-9. doi: 10.5005/jp-journals-10005-1260. Epub 2015 Feb 9. PMID 25709297
- [Background] Ramos-Jorge ML, Ramos-Jorge J, Vieira de Andrade RG, Marques LS. Impact of exposure to positive images on dental anxiety among children: a controlled trial. Eur Arch Paediatr Dent. 2011 Aug;12(4):195-9. doi: 10.1007/BF03262806. PMID 21806903
- [Background] Malhotra R, Gandhi K, Kumar D, Ahuja S, Kapoor R, Sahni A. A Comparative Study to evaluate Parent's Ability to assess Dental Fear in their 6- to 10-year-old Children using Children's Fear Survey Schedule-Dental Subscale. Int J Clin Pediatr Dent. 2018 May-Jun;11(3):205-209. doi: 10.5005/jp-journals-10005-1512. Epub 2018 Jun 1. PMID 30131642
- [Background] Venham LL, Gaulin-Kremer E. A self-report measure of situational anxiety for young children. Pediatr Dent. 1979 Jun;1(2):91-6. No abstract available. PMID 399677